CLINICAL TRIAL: NCT00004061
Title: A Randomized Double-Blind, Placebo-Controlled Trial of Recombinant Human Keratinocyte Growth Factor (rHuKGF) in Patients With Hematologic Malignancies Undergoing Total Body Irradiation (TBI) and High-Dose Chemotherapy With Autologous Peripheral Blood
Brief Title: Biological Therapy in Treating Patients Undergoing Radiation Therapy, Chemotherapy, and Peripheral Stem Cell Transplantation for Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: AMGEN-KGF-980231-04; MSKCC-99029; CDR0000067261 (Registry Identifier: PDQ (Physician Data Query)); NCI-G99-1574
Record Dates: First submitted 1999-12-10; First posted 2004-05-25 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2009-12

CONDITIONS: Leukemia; Lymphoma; Oral Complications
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; oral complications; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; secondary acute myeloid leukemia; stage I mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone | interventions — Filgrastim; Fibroblast Growth Factor 7; Cyclophosphamide; Etoposide; Ifosfamide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Biological: palifermin
Drug: cyclophosphamide
Drug: etoposide
Drug: ifosfamide
Procedure: peripheral blood stem cell transplantation
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Biological therapy using growth factors may be effective in reducing side effects in patients who have hematologic cancer and are receiving radiation therapy, chemotherapy, and peripheral stem cell transplantation.

PURPOSE: Randomized phase II trial to study the effectiveness of biological therapy to reduce side effects in patients who are undergoing radiation therapy, chemotherapy, and peripheral stem cell transplantation in treating lymphoma or leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of recombinant human keratinocyte growth factor (rHuKGF) in reducing severe oral mucositis induced by total body irradiation and high dose chemotherapy in patients with hematologic malignancies. II. Compare the incidence of severe oral mucositis, the use of transdermal or perenteral opioid analgesics, and the incidence and duration of grade 2-4 diarrhea with or without rHuKGF in these patients. III. Determine the quality of life of these patients. IV. Determine the duration of febrile neutropenia and the duration of treatment with intravenous antifungals or antibiotics in these patients.

OUTLINE: This is a randomized, double blind, placebo controlled, multicenter study. Patients are stratified according to center. Patients are randomized to one of three treatment arms. Arm I: Patients receive recombinant human keratinocyte growth factor (rHuKGF) IV on days -11 to -9, -5, and 0 to 2. Total body irradiation (TBI) is administered twice a day on days -8 to -5. Patients receive etoposide IV over 4 hours on day -4 and cyclophosphamide IV over 1 hour on day -2 (some patients may receive an alternate regimen of ifosfamide IV over 1 hour on days-4 to 0 followed each day by etoposide IV over 23 hours). Filgrastim (G-CSF) is administered subcutaneously (SQ) beginning on day 0 and continuing for up to 21 days until blood counts recover. Autologous peripheral blood stem cells (PBSC) are infused on day 0. Arm II: Patients receive rHuKGF on days -11 to -9 and -5 as in arm I. Placebo is administered on days 0 to 2. TBI, chemotherapy, and PBSC transplantation are administered as in arm I. Arm III: Patients receive placebo on days -11 to -9, -5, and 0 to 2. TBI, chemotherapy, and PBSC transplantation are administered as in arm I. Quality of life is assessed prior to treatment, daily during therapy and until day 28 after transplantation. Patients are followed at day 28 and approximately day 60-100.

PROJECTED ACCRUAL: At least 111 patients (37 per arm) will be accrued for this study within 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of one of the following: Non-Hodgkin's lymphoma Hodgkin's disease Acute myelogenous leukemia Acute lymphoblastic leukemia Chronic myelogenous leukemia Chronic lymphocytic leukemia Eligible for fractionated total body irradiation plus high dose chemotherapy followed by autologous peripheral blood stem cell support No prior entry into this study

PATIENT CHARACTERISTICS: Age: 18 to 65 Performance status: Karnofsky 70-100% SWOG 0 or 1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count greater than 1,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL Renal: Creatinine no greater than 2 mg/dL Cardiovascular: No New York Heart Association class III or IV heart disease Pulmonary: DLCO at least 60% predicted Other: No other prior or concurrent malignancy No active infection or oral mucositis No diabetes mellitus requiring insulin HIV negative No sensitivity to E. coli derived products Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No prior bone marrow or peripheral blood stem cell transplantation No concurrent interleukin-11 Chemotherapy: See Disease Characteristics No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior extensive radiotherapy that would preclude study irradiation Surgery: Not specified Other: At least 30 days since prior investigational study No other concurrent investigational agents No concurrent prophylactic oral cryotherapy during study chemotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 1999-05; Primary Completion 2003-05 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric W. Hedrick, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States